

#### NON-INTERVENTIONAL STATISTICAL ANALYSIS PLAN FOR SECONDARY DATA COLLECTION STUDY



# Non-Interventional Study Protocol < 80661181>

# Safety and effectiveness of apixaban in very elderly patients with NVAF compared to warfarin using administrative claims data

Statistical Analysis Plan(SAP)

Version: Ver.2.0

Author: PPD Pfizer Japan

Date: 10-Aug-2023

# **TABLE OF CONTENTS**

| 1. | AMENDMENTS FROM PREVIOUS VERSION(S) | 4 |
|---|---|---|
| 2. | INTRODUCTION | 4 |
| 2 | STUDY DESIGN | 6<br>6<br>7 |
| 3. | HYPOTHESES AND DECISION RULES | 7 |
| 3.1<br>3.2 | STATISTICAL DECISION RULES | 7 |
| 4. | ANALYSIS SETS/POPULATIONS | 7 |
| 4.2<br>4.3 | 4.1.1. Inclusion criteria | 7<br>8<br><b>8</b> |
| 4.5 | SAMPLE SIZE CALCULATION | 9 |
| 5. | ENDPOINTS AND COVARIATES | |
| 5.1<br>5.2<br>5.2 | EFFICACY/EFFECTIVENESS ENDPOINT(S) 5.1.1. Primary effectiveness endpoint and primary analyses 5.1.2. Secondary effectiveness endpoint and secondary analyses SAFETY ENDPOINTS 5.2.1. Primary safety endpoint and primary analyses 5.2.2. Secondary safety endpoint and secondary analyses OTHER ENDPOINTS | <b>11</b><br>11<br><b>11</b><br><b>11</b><br>12 |
| 5.1<br>5.2<br>5.3 | EFFICACY/EFFECTIVENESS ENDPOINT(S) 5.1.1. Primary effectiveness endpoint and primary analyses 5.1.2. Secondary effectiveness endpoint and secondary analyses SAFETY ENDPOINTS | 11<br>11<br>11<br>11<br>12<br>12 |
| 5.1<br>5.2<br>5.3<br>5.4 | EFFICACY/EFFECTIVENESS ENDPOINT(S) 5.1.1. Primary effectiveness endpoint and primary analyses 5.1.2. Secondary effectiveness endpoint and secondary analyses SAFETY ENDPOINTS 5.2.1. Primary safety endpoint and primary analyses 5.2.2. Secondary safety endpoint and secondary analyses OTHER ENDPOINTS COVARIATES | 11<br>11<br>11<br>11<br>12<br>12 |

| 7.2.1. | Safety Analysis | 19 |
|----------|-----------------------------------------------------------|----|
| 7.2.2. | Analysis of Efficacy Analysis | |
| 7.2.3. | Sensitivity analysis | 19 |
| 7.2.4. | Summary of Analyses | 20 |
| 8. LIST | OF TABLES AND TABLE SHELLS | 23 |
| 9. REFI | ERENCES | 23 |
| 10. APP | ENDICES | 23 |
| 10.1. AP | PENDIX 1: DATA DERIVATION DETAILS | 23 |
| | PENDIX 2: ADDITIONAL STATISTICAL METHODOLOGY DETAILS | |
| | PENDIX 3: DIAGNOSIS AND PROCEDURE CODES USED IN THE STUDY | |
| | List of diagnosis code | |
| | List of procedure code | |
| 10.3.3. | Stroke related medical history | 40 |
| 10.3.4. | | 40 |
| 10 3 5 | other codes | 16 |

#### 1. AMENDMENTS FROM PREVIOUS VERSION(S)

From version 1.0 to version 1.1, no substantial changes have been made and only asministrative changes including correction of typos as follows; 1) in SCI

2) in 7.2.4 Summary of analysis, "time course of proportion of stroke-free" was changed to "time course of proportion of stroke/SE-free". Both changes are considered to be just administrative ones and little impact on the results would be expected.

From version 1.1 to version 2.0, two major changes have been made. Firstly, patient registration period descried in the section 2.1.1 was changed from "2008 to 2021" to "February 26, 2013 to December 31, 2021" to consider the launch date of apixaban in Japan. This change will make concurrent active control (i.e., warfarin cohort) for apixaban cohort. Secondly, calculation of propensity score was modified in the section "7.1.2.1" to adjust effect of time on treament selection (i.e., warfarin or apixaban). Propensity scores will be calculated by calendar year of index date.

#### 2. INTRODUCTION

The number of patients with atrial fibrillation (AF) has been in the elderly patients has been increasing worldwide[1]. Especially, Japan is a very elderly society compared to other countries in Europe and the United States, and there are many very elderly patients with NVAF who are treated with any of anticoagulant and there are considerable number of patients who are newly diagnosed with NVAF even in their 80's and 90's. In the previous real-world database study conducted in Japan (CER3 study), the mean age of patients with non-valvular AF (NVAF) were 75-78 years old[2]. Most of these very elderly people have many complications, including severe ones, and take many medications chronically. In addition, many elderly patients have low body weight, sarcopenia, low ADL, frailty or frail-like characteristics, or high risk of falls. There has been much debate and inconclusive evidence on the value of anticoagulation for these very elderly patients with NVAF[1, 3, 4,].

ARISTOTLE study has shown that apixaban is superior or equivalent to warfarin in various populations including populations at higher risk. However, there are few studies in the real-world settings regarding very elderly patients who are at higher risk.

Research question and objectives:

The ARISTOTLE study and various real-world evidence (RWE) have shown that apixaban is superior or equivalent to warfarin in safety and effectiveness profile. Subgroup analyses of the ARISTOTLE study suggested that superiority over warfarin could be consistent in most populations including high risk populations. Study hypothesis and clinical questions in this study is apixaban is superior to warfarin in both safety and effectiveness even in the very elderly patients with NVAF in the real-world settings.

The clinical question of this study is that apixaban has a superior effectiveness and safety profile compared to warfarin, even in very elderly patients who are at particularly high risk, such as those with CCI , frail or frail patients, those with significant comorbidities, those with polypharmacy, and those at high risk of falls.

The objective of this study is to investigate safety and effectiveness of apixaban compared to warfarin in very elderly patients with NVAF.

## 2.1. STUDY DESIGN

This is a retrospective non-intervention observational study to evaluate the difference in safety and effectiveness between apixaban and warfarin using a database provided by Medical Data Vision Co. Ltd. (MDV Co. Ltd.). Eligible patients will be extracted from the database and allocated to the pre-defined cohorts based on the actual age, age of NVAF diagnosis and types of anticoagulant therapy.

Based on the age category and anticoagulants on the index date (a date when patients initiated an anticoagulant for prevention of stroke/SE), eligible patients will be allocated to some cohorts. Patient characteristics will be balanced by an Inverse probability of treatment weighting (IPTW) method, and risk of stroke/SE (primary effectiveness endpoint) and major bleeding (primary safety endpoint) will be compared. Hazard ratios and 95% confident intervals will be calculated by using a Cox proportional hazard method with a robust sandwich variance estimator to account for induced correlations among weighted patients.

#### 2.1.1. Study population

Patients registered in the MDV database from February 26, 2013 to December 31, 2021 will be used. First, patients with a NVAF diagnosis and received apixaban or warfarin as an anticoagulant after the NVAF diagnosis will be identified and then among them only patients who are 80 or older when they initiated these medications.

Based on the first anticoagulant prescribed, eligible patients will be allocated to one of two cohorts, an apixaban or warfarin cohort. Comparison will be made between these cohorts after balancing of the patient characteristics by a IPTW with stabilized weights (s-IPTW) method.



#### 2.1.2. Data source

Medical Data Vision database, commercially available administrative claims database from hospitals introducing DPC (Diagnosis Procedure Combination) system, which comprises administrative data pertaining to approximately 39 million individuals (as of 2021 Dec.) managed in the inpatient and outpatient settings. In this database, all patients have been de-identified and no personal information resulting the identification of individuals.

#### 2.1.3. Treatment/cohort labels

- Apixaban cohort: patients diagnosed with non-valvular atrial fibrillation who are 80 or older when they initiated apixaban as an anticoagulant.
- 2. <u>Warfarin cohort:</u> patients diagnosed with non-valvular atrial fibrillation who are 80 or older when they initiated warfarin as an anticoagulant.

#### 2.2. STUDY OBJECTIVES

The objective of this study is to investigate safety and effectiveness of apixaban compared to warfarin in very elderly patients with NVAF.

The purposes of this study are 1) to characterize the primary and secondary prevention patients, 2) incidence rates of stroke/SE or major bleeding in each cohort and 3) is to investigate for Japanese secondary prevention patients as RWE on the effectiveness and safety of apixaban compared to warfarin in patients with NVAF.

#### 3. HYPOTHESES AND DECISION RULES

#### 3.1. STATISTICAL HYPOTHESES

Not applicable

#### 3.2. STATISTICAL DECISION RULES

When the effect of factors in an analysis is statistically evaluated, the alpha level of 0.05 will be referred.

#### 4. ANALYSIS SETS/POPULATIONS

#### 4.1. FULL ANALYSIS SET

#### 4.1.1. Inclusion criteria

Patients must meet all the following inclusion criteria to be eligible for inclusion in the study.

1. Diagnosed with AF anytime in the baseline period or on the index date, also have definitive diagnosis of AF anytime in the baseline period, on the index date, or post-index period.

- 2. Prescribed apixaban or warfarin on or after the day of AF diagnosis. The first observed prescription will be used to identify the patient's index date and treatment cohort
- 3. No use of the any OACs during the baseline period (the 180 days before the index date)
- 4. Age of 18 years or older on the index date.
- 5. Index date is at age 80 or older

#### 4.1.2. Exclusion criteria

Patients meeting any of the following criteria will not be included in the study:

- Having a diagnosis of valvular atrial fibrillation, post-operative atrial fibrillation, rheumatic atrial fibrillation or mechanical-valvular atrial fibrillation during the baseline and postindex period
- 2. Having a cardiac surgery procedure record during the baseline period
- 3. Having a joint replacement procedure record during the baseline period
- 4. Having a procedure of prosthetic heart valve during the baseline period
- 5. Having a diagnosis of venous thromboembolism during the baseline period
- 6. Female patients with pregnancy during the follow-up period
- 7. Patients prescribed "off-label" doses of OACs (per Japanese package insert of each OAC) or patients treated with OAC but in "off-label" or "contraindicated" manners.

#### 4.2. SAFETY ANALYSIS SET

Bleeding other than safety-related reactions will not be investigated here. Bleeding events will be evaluated using the same analysis set as effectiveness.

#### 4.3. OTHER ANALYSIS SET

Not applicable. All eligible patients will be used for the analysis except the pre-designated subanalysis.





#### 4.5. SAMPLE SIZE CALCULATION

This study is a retrospective analysis of the structured data in the database and all eligible patients will be used for analysis.

The results of the feasibility assessment are shown below,

Table 1. The number of patients

| Patient group | Number of patients |
|---|---|
| Patients diagnosed with NVAF at 80 years or an age older than 80 and data when patients are 80 or older are available. | |
| Treated with apixaban | 76,260 |
| Treated with warfarin | 62,453 |


Note that not all of these patients are eligible for this study because no inclusion and exclusion criteria were applied when the number of patients was estimated.

In the previous study (CER3)[2], incidence rate of major bleeding and stroke/SE were 2.5% for warfarin and 1.18 % for apixaban and 1.92% for warfarin and 0.98% for apixaban, respectively. Hazard ratios for major bleeding and stroke/SE were 0.58 and 0.57, respectively. In CER3 subgroup analysis on age, hazard ratios in sub-cohort of ages ≥ 80 years were 0.59 and 0.53 for major bleeding and stroke/SE, respectively. Although populations used for analysis are different (in the CER3 study, warfarin and apixaban could be started at any age, whereas in this study, the starting date for warfarin and apixaban was restricted to ages 80 years and older), difference may not be very large because the mean age of populations in CER3 is around 77 years old in both warfarin and apixaban cohorts. Sample size calculation was performed based on the CER3 results of older age subgroup analysis.

Table 2. Sample size calculation

| Type I error rate 0.05 Type II error rate 0.2 Hazard ratio 0.59 N ratio in apixaban and 1:1 warfarin cohorts Event rate for warfarin 2.5%/year Event rate for apixaban 1.18%/year Total events needed 113 Estimated number of patients 6,141 |
|---|
| Type I error rate 0.05 Type II error rate 0.2 Hazard ratio 0.59 N ratio in apixaban and 1:1 warfarin cohorts Event rate for warfarin 2.5%/year Event rate for apixaban 1.18%/year Total events needed 113 |
| Type II error rate 0.2 Hazard ratio 0.59 N ratio in apixaban and 1:1 warfarin cohorts Event rate for warfarin 2.5%/year Event rate for apixaban 1.18%/year Total events needed 113 |
| Hazard ratio 0.59 N ratio in apixaban and 1:1 warfarin cohorts Event rate for warfarin 2.5%/year Event rate for apixaban 1.18%/year Total events needed 113 |
| N ratio in apixaban and warfarin cohorts Event rate for warfarin Event rate for apixaban Total events needed 1:1 2.5%/year 1.18%/year 113 |
| warfarin cohorts Event rate for warfarin Event rate for apixaban Total events needed 2.5%/year 1.18%/year 113 |
| Event rate for apixaban 1.18%/year Total events needed 1.18%/year |
| Total events needed 113 |
| Estimated number of patients 6,141 |
| For Stroke/SE |
| Type I error rate 0.05 |
| Type II error rate 0.2 |
| Hazard ratio 0.53 |
| N ratio in apixaban and 1:1 warfarin cohorts |
| Event rate for warfarin 1.92%/year |
| Event rate for apixaban 0.98%/year |
| Total events needed 78 |
| Estimated number of patients 5,379 |

Even allowing for the fact that 1) event rate may be higher because only patients whose index date is at 80 years or older (that is, high risk population for both stroke/SE and major PFIZER CONFIDENTIAL

bleeding) and 2) not all of patients in Table 1 above are eligible for this study, the number of eligible patients could be enough for primary safety and effectiveness analyses with appropriate statistical power.

#### 5. ENDPOINTS AND COVARIATES

#### 5.1. EFFICACY/EFFECTIVENESS ENDPOINT(S)

#### 5.1.1. Primary effectiveness endpoint and primary analyses

Primary effectiveness endpoint is incidence of a composite of Stroke/SE ("cardiogenic cerebral embolism", "cerebral infarction", hemorrhargic stroke or SE) in NVAF patients treated with warfarin or apixaban. TIA is not included in the outcome (not regarded as stroke).

- 1. Incidence of stroke/SE (per 1,000 person-year)
- Survival curves of stroke/SE-free patients (Kaplan-Meier curves) will be drawn for apixaban and warfarin cohorts. Difference in the two curves will be evaluated by a Logrank test.

Risk of stroke/SE in each cohort will be compared between balanced warfarin and balanced apixaban cohorts by using Cox proportional hazard analysis. Hazard ratio with 95% confident intervals will be calculated.

#### 5.1.2. Secondary effectiveness endpoint and secondary analyses

Secondary effectiveness endpoints are the incidence of "cardiogenic cerebral embolism" or "ischemic stroke" during the follow-up period in NVAF patients treated with warfarin or apixaban.

For each secondary endpoint, like the primary analysis, incidence of the secondary endpoint, Kaplan Meier curves and Hazard ratios with 95% confident intervals will be calculated

#### 5.2. SAFETY ENDPOINTS

#### 5.2.1. Primary safety endpoint and primary analyses

Primary safety endpoint is incidence of major bleeding, which is defined as any bleeding requiring hospitalization.

1. Incidence of Major bleeding (per 1,000 person-year)

- Survival curves of major bleeding-free patients (Kaplan-Meier curves) will be drawn for apixaban and warfarin cohorts. Difference in the two curves will be evaluated by a Logrank test.
- 3. Risk of major bleeding in each cohort will be compared between balanced warfarin and balanced apixaban cohorts by using Cox proportional hazard analysis. Hazard ratio with 95% confident intervals will be calculated.

#### 5.2.2. Secondary safety endpoint and secondary analyses

Secondary safety endpoints are the incidence of "intracranial hemorrhage", "gastrointestinal bleeding" or "intraocular bleeding" during the follow-up period in NVAF patients treated with warfarin or apixaban.

For each secondary endpoint ("intracranial hemorrhage", "gastrointestinal bleeding" or "intraocular bleeding"), like the primary analysis, incidence of each secondary endpoint, Kaplan-Meier curves and Hazard ratios with 95% confident intervals will be calculated

#### 5.3. OTHER ENDPOINTS

None

#### **5.4. COVARIATES**

| Items | definitions | roles |
|---|---|---|
| Gender | Male or female | Patient characteristics |
| | | CCI |
| Body weight | ≥ 60 kg or < 60 kg | Patient characteristics |
| eGFR (continuous) | Value in the baseline If a patient has multiple eGFR values, the values closest to the index date will be adopted | Patient<br>characteristics |
| eGFR (categorical) | ≥ 50 ml/min or < 50 ml/min | Patient characteristics |
| Serum creatinine (continuous) | Value in the baseline If a patient has multiple eGFR values, the values closest to the index date will be adopted | Patient<br>characteristics |

| Serum creatinine (categorical) | ≥ 1.5mg/mL or < 1.5<br>mg/mL | Patient characteristics |
|---|---|---|
| CHADS2 | CHADS2 score will<br>be calculated based<br>on age and the<br>presence of<br>congestive heart<br>failure, hypertension,<br>diabetes, and stroke<br>or TIA. | Patient<br>characteristics |
| CHA2DS2-VASc | CHA2DS2-VASc<br>score will be<br>calculated based on<br>age and the<br>presence of<br>congestive heart<br>failure, hypertension,<br>diabetes, stroke or<br>TIA, vascular disease<br>and sex category. | Patient<br>characteristics |
| CCI | | |

Medications Defined using prespecified drug-Patient Treated with antiplatelet drug in baseline specific codes: Yes characteristics or No

Defined usina prespecified drug-Patient Treated with NSAIDs in baseline specific codes: Yes characteristics or No Defined using prespecified drug-Treated with gastric secretion inhibitor in Patient specific codes: Yes baseline characteristics or No Defined using prespecified drug-Patient Treated with statin-based drug in baseline specific codes: Yes characteristics or No Defined using prespecified drug-Patient Treated with anti-hypertensives in baseline specific codes: Yes characteristics or No Defined using prespecified drug-Patient Treated with anti-arrhythmics in baseline specific codes: Yes characteristics or No Defined using prespecified drug-Patient Treated with beta-blockers in baseline specific codes: Yes characteristics or No **Procedures** Defined using prespecified medical Patient Cardioversion procedure codes: characteristics Yes or No Defined using prespecified medical Patient Cardiac ablation procedure codes: characteristics Yes or No **Anticogulation** INR (warfarin cohort) Continuous variable. Patient \* Only available for characteristics patients treated with warfarin 2.5 mg BID or 5mg Patient Apixaban doses BID \* Only available characteristics

Chronically prescribed medicines

Medicines that had been prescribed at least for 30 days during the baseline period.

for patients treated with apixaban

#### 6. HANDLING OF MISSING VALUES

No imputation for missing values will be conducted.

#### 7. STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES

#### 7.1. STATISTICAL METHODS

#### 7.1.1. Patient characteristics

Means with standard deviations or medians with quartile values (25% and 75% values) will be provided for continuous variables when performing descriptive analysis of continuous data. Numbers and percentages will be provided for dichotomous and polychotomous variables when performing descriptive analysis of categorical data. Bivariate comparisons of baseline characteristics and outcomes measures will be provided. Appropriate tests (unpaired t-test or Mann-Whitney U-test, categorical variables: Chi-square or Fisher's exact test) will be used based on the distribution of the measure.

#### 7.1.2. Patient characteristics balancing

In this study, cohorts with balanced patient characteristics (s-IPTW warfarin cohort and s-IPTW apixaban cohort) will be created from raw cohorts (raw warfarin and raw apixaban cohorts). A propensity score will be calculated based on multivariable logistic regressions in order to account for confounding effects and to ensure that patient characteristics will be balanced between the warfarin cohort and apixaban cohort. An inverse probability of treatment weighting (IPTW) method using the calculated propensity score will be applied. To avoid sample size inflation and to ensure appropriate estimation of variances, s-IPTW (stabilized IPTW) will be used here.

#### 7.1.2.1. Calculation of propensity score

Propensity scores will be estimated by calendar year of index date based on multivariable logistic regression analyses that incorporate potential predictors of therapy as independent variables in the regression and cohort status (prescription of warfarin or apixaban) as the outcome. Consecutive calendar years of index dates may be collapsed to build logistic regression model with robustness. The following covariates will be included in the logistic regression:

- age on index date
- age at NVAF diagnosis
- gender

- CHADS<sub>2</sub> score in baseline
- CHA<sub>2</sub>DS<sub>2</sub>-VASc score in baseline
- heart failure diagnosis in baseline
- coronary heart disease diagnosis in baseline
- peripheral arterial disorder diagnosis in baseline
- myocardial infarction diagnosis in baseline
- hyperthyroidism or thyrotoxicosis in baseline
- TIA diagnosis in baseline
- stroke or SE diagnosis in baseline
- renal dysfunction diagnosis in baseline
- liver dysfunction diagnosis in baseline
- bleeding diagnosis in baseline
- hypertension diagnosis in baseline
- diabetes mellitus diagnosis in baseline
- treated with antiplatelet drug in baseline
- treated with NSAIDs in baseline
- treated with gastric secretion inhibitor in baseline
- treated with statin-based drug in baseline
- treated with anti-hypertensives in baseline
- treated with anti-arrhythmics in baseline
- treated with beta-blockers in baseline
- treated with heparins in baseline
- cardioversion in baseline

#### 7.1.2.2. IPTW with stabilized weights[6]

IPTW with stabilized weights will be used to balance patient characteristics between two groups using propensity score calculated by using a multivariable logistic model as mentioned above (see above 7.1.2.1). However, if a treated patient has a very low propensity score, a very large weight can be created. Large weights can increase the variability of estimated treatment effect. In order to address this, the weights can be stabilized. Stabilized weights will be calculated by using a formula shown below, by multiplying the treatment and control weights by a constant, equal to the expected value of being in the treatment or comparison cohorts, respectively.

$$W_i = \frac{Z}{PS_i} + \frac{1-Z}{1-PS_i}$$
, z: probability of treatment without considering covariates

The distribution of the stabilized weight will be reviewed. If there are extreme outliers, the large weights could be set to a less extreme value (e.g. recoding all weights that are outside 5th and 95th percentile). If needed, truncation can be done after stabilizing the weights. After the weights are applied, the balance of the baseline covariates will be assessed. First, the means and proportions of baseline variables are compared. The standardized difference compares the difference in means in units of the standard deviation. If the standardized difference is less than 10%, the covariates are considered balanced.

#### 7.1.2.3. Calculation of event rate

Patients who experience a clinical endpoint event after the earlier of their discontinuation of the index OAC, switching from the index OAC, withdrawal from the database, or the end of intended follow-up period will be censored. Patients who do not experience a clinical endpoint event will be censored at the earlier of their discontinuation of the index OAC, switching from the index OAC or withdrawal from the database will be censored.

Using the number of patients who experience each endpoints and the total observation period, incidence rate of each endpoint will be calculated and be presented as per 1,000 person-years.

#### 7.1.2.4. Kaplan-Meier Method

For each endpoint, Kaplan-Meier curves will be plotted for the time from the index date to first event by index OAC treatment in each of the IPTW cohorts. The log-rank test is used for comparison between two curves.

#### 7.1.2.5. Calculation of hazard ratio with 95% confident intervals

Cox proportional hazards model will be used to compare endpoints in each of the sIPTW cohorts, with robust sandwich estimates to account for the clustering within balanced sets. The Cox proportional hazards model will include only index OAC treatment (apixaban or warfarin) as the independent variable if patient characteristics are well balanced between groups based on standardized difference in components of the PS. If not balanced, the unbalanced variable will be also included to the model in addition to the index OAC treatment. The hazard ratios with corresponding 95% confidence intervals and p-values will be reported.



#### 7.2. STATISTICAL ANALYSIS

#### 7.2.1. Safety Analysis

This is a database study and safety analyses will not be performed because it is not possible to identify adverse events directly caused by the drug or suspected to be related to the drug. Only incidence of major bleeding, occurred during the follow-up periods, will be compared between s-IPTW apixaban and warfarin cohorts. See 5.2.1 and 7.1 above.

#### 7.2.2. Analysis of Efficacy Analysis

See 7.1 above

#### 7.2.3. Sensitivity analysis

E-values will be calculated to assess the extent of unmeasured confounding on findings from primary analyses of effectiveness and safety outcomes. E-value is a measure developed by VanderWeele and Ding (2017) as the minimal strength of association between a hypothetical unmeasured confounder with both the treatment and outcome to explain away the identified association between treatment and the outcome.

# 7.2.4. Summary of Analyses

| Outcome | Analysis<br>Set | Endpoint | Subgroup | Statistical Method | Covariates/Strata | Missing Data |
|---|---|---|---|---|---|---|
| Incidence rate of stroke/SE | Balanced cohorts | Primary<br>effectiveness | None | 1000 person-years | Refer to 5.1.1 | No imputation |
| Incidence of cardiogenic cerebral embolism | Balanced cohorts | Secondary<br>effectiveness | None | 1000 person-years | Refer to 5.1.2 | No imputation |
| Incidence of cerebral infarction | Balanced cohorts | Secondary<br>effectiveness | None | 1000 person-years | Refer to 5.1.2 | No imputation |
| Incidence rate of major bleeding | Balanced cohorts | Primary safety | None | 1000 person-years | Refer to 5.2.1 | No imputation |
| Incidence rate of intracranial hemorrhage | Balanced cohorts | Secondary safety | None | 1000 person-years | Refer to 5.2.2 | No imputation |
| Incidence rate of gastrointestinal bleeding | Balanced cohorts | Secondary<br>safety | None | 1000 person-years | Refer to 5.2.2 | No imputation |
| Incidence of rate of intraocular bleeding | Balanced cohorts | Secondary<br>safety | None | 1000 person-years | Refer to 5.2.2 | No imputation |
| Time course of proportion of stroke/SE -free NVAF patients | Balanced cohorts | Primary effectiveness | None | Kaplan-Meier curves | Refer to 5.1.1 | No imputation |
| Time course of proportion of cardiogenic cerebral embolism-free NVAF patients | Balanced cohorts | Secondary<br>effectiveness | None | Kaplan-Meier curves | Refer to 5.1.2 | No imputation |
| Time course of proportion of cerebral infarction"-free NVAF patients | Balanced cohorts | Secondary<br>effectiveness | None | Kaplan-Meier curves | Refer to 5.1.2 | No imputation |

| Time course of proportion of major bleeding-<br>free NVAF patients | Balanced cohorts | Primary safety | None | Kaplan-Meier curves | Refer to 5.2.1 | No imputation |
|---|---|---|---|---|---|---|
| Time course of proportion of intracranial hemorrhage-free NVAF patients | Balanced cohorts | Secondary<br>safety | None | Kaplan-Meier curves | Refer to section 5.2.2 | No imputation |
| Time course of proportion of gastrointestinal bleeding-free NVAF patients | Balanced cohorts | Secondary<br>safety | None | Kaplan-Meier curves | Refer to section 5.2.2 | No imputation |
| Time course of proportion of intraocular bleeding-free NVAF patients | Balanced cohorts | Secondary<br>safety | None | Kaplan-Meier curves | Refer to section 5.2.2 | No imputation |
| Risk of stroke/SE during the follow-up period in NVAF patients (Hazard ratio, apixaban versus warfarin) | Balanced cohorts | Primary<br>endpoint | None | Cox proportional hazards regression model | Refer to 5.1.1 | No imputation |
| Risk of cardioembolic stroke during the follow-up period in NVAF patients (Hazard ratio, apixaban versus warfarin) | Balanced cohorts | Secondary<br>effectiveness | None | Cox proportional hazards regression model | Refer to 5.1.2 | No imputation |
| Risk of cerebral infarction during the follow-<br>up period in NVAF patients (Hazard ratio,<br>apixaban versus warfarin) | Balanced cohorts | Secondary<br>effectiveness | None | Cox proportional hazards regression model | Refer to 5.1.2 | No imputation |
| Risk of major bleeding during the follow-up period in NVAF patients (Hazard ratio, apixaban versus warfarin) | Balanced cohorts | Primary safety | None | Cox proportional hazards regression model | Refer to 5.2.1 | No imputation |
| Risk of intracranial hemorrhage during the follow-up period in NVAF patients (Hazard ratio, apixaban versus warfarin) | Balanced cohorts | Secondary<br>safety | None | Cox proportional hazards regression model | Refer to 5.2.2 | No imputation |
| Risk of gastrointestinal tract bleeding during the follow-up period in NVAF patients (Hazard ratio, apixaban versus warfarin) | Balanced cohorts | Secondary<br>safety | None | Cox proportional hazards regression model | Refer to 5.2.2 | No imputation |

NIS Protocol <B0661181>

# Statistical Analysis Plan

| Risk of intraocular bleeding during the follow-up period in NVAF patients (Hazard ratio, apixaban versus warfarin) | Balanced cohorts | Secondary<br>safety | None | Cox proportional hazards regression model | Refer to 5.2.2 | No imputation |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

#### 8. LIST OF TABLES AND TABLE SHELLS

None

#### 9. REFERENCES

- 1. Bauersachs, R.M. and J. Herold, *Oral Anticoagulation in the Elderly and Frail.* Hamostaseologie, 2020. **40**(1): p. 74-83.
- 2. Kohsaka, S., et al., Safety and effectiveness of non-vitamin K oral anticoagulants versus warfarin in real-world patients with non-valvular atrial fibrillation: a retrospective analysis of contemporary Japanese administrative claims data. Open Heart, 2020. **7**(1): p. e001232.
- 3. Patti, G., et al., Thromboembolic Risk, Bleeding Outcomes and Effect of Different Antithrombotic Strategies in Very Elderly Patients With Atrial Fibrillation: A Sub-Analysis From the PREFER in AF (PREvention of Thromboembolic Events-European Registry in Atrial Fibrillation). J Am Heart Assoc, 2017. 6(7).
- 4. Chao, T.F., et al., *Oral anticoagulants in extremely-high-risk, very elderly (>90 years) patients with atrial fibrillation*. Heart Rhythm, 2021. **18**(6): p. 871-877.
- 5. Granger, C.B., et al., *Apixaban versus warfarin in patients with atrial fibrillation.* N Engl J Med, 2011. **365**(11): p. 981-92.
- 6. Xu, S., et al., Use of stabilized inverse propensity scores as weights to directly estimate relative risk and its confidence intervals. Value Health, 2010. **13**(2): p. 273-7.

#### 10. APPENDICES

#### 10.1. APPENDIX 1: DATA DERIVATION DETAILS

Not applicable

#### 10.2. APPENDIX 2: ADDITIONAL STATISTICAL METHODOLOGY DETAILS

Not applicable

# 10.3. APPENDIX 3: DIAGNOSIS AND PROCEDURE CODES USED IN THE STUDY

### 10.3.1. List of diagnosis code

| Variable Used in Study | ICD-10<br>Code <sup>*</sup> | Additional rules on Data Extraction |
|---|---|---|
| Atrial fibrillation | 148 | |
| Post-operative atrial fibrillation | 8847772 | Standard disease code |
| Valvular atrial fibrillation | 8846941 | Standard disease code |

| Variable Used<br>in Study | ICD-10<br>Code* | Additional rules on Data Extraction |
|---|---|---|
| Rheumatic atrial fibrillation | 105 | |
| | 106 | |
| | 107 | |
| | 108 | |
| | 109 | |
| Mechanical-valvular atrial fibrillation | T820 | |
| Hyperthyroidism or thyrotoxicosis | E05 | |
| Heart failure | I110 | |
| | 1500 | |
| | I501 | Exclude cardiac asthma |
| | 1509 | |
| Hypertension | H208 | Include only hypertensive iridocyclitis |
| | H350 | Include only hypertensive retinopathy and hypertensive neuroretinopathy |
| | I10 | |
| | I110 | |
| | I119 | |
| | I120 | |
| | I129 | Include only hypertensive renal disease, hypertensive nephropathy and hypertensive nephrosclerosis |
| | I139 | |
| | I150 | |
| | I151 | |
| | I152 | |
| | I158 | |
| | I159 | |
| | I619 | Include only hypertensive intracerebral hemorrhage |
| | 1674 | |
| Diabetes | E10 | |
| | E11 | |
| | E12 | |
| | E13 | |
| | E14 | |
| Hemorrhage stroke | 160 | |
| | l61 | |
| | 162 | Exclude non-traumatic extradural haemorrhage |

| Variable Used in Study | ICD-10<br>Code* | Additional rules on Data Extraction |
|---|---|---|
| Ischemic stroke | 163 | On Data Extraorion |
| | 3489032 | standard disease code |
| | 4371003 | |
| | 4379014 | |
| | 3448002 | |
| | 3448028 | |
| | 3489029 | |
| | 3489035 | |
| | 4379006 | |
| TIA | H340 | |
| | G450 | |
| | G451 | |
| | G458 | |
| | G459 | |
| Systemic embolism | 1740 | Include only abdominal aortic embolism |
| | 1741 | Include only aortic embolism |
| | 1742 | Include only acute arterial occlusive disease of arteries of upper extremities |
| | 1743 | Include only femoral arterial occlusion and acute arterial occlusive disease of arteries of lower extremities |
| | 1744 | |
| | 1745 | Include only iliac artery embolism |
| | 1748 | Include only hepatic artery embolism |
| | 1749 | Include only thromboembolism, embolic infarction, aortic embolism |
| Peripheral vascular disorder | 1702 | Include only atherosclerosis and arteriosclerosis obliterans |
| | 1709 | |
| | 1731 | Include only Buerger's disease |
| | 1739 | Exclude peripheral circulatory failure, cerebrovascular spasm, and angiospasm pf the extremities |
| | 1742 | |
| | 1743 | |
| | 1745 | |
| | 1748 | Include only subclavian artery stenosis |
| Aortic plaque | 4400011 | Standard disease code |
| | 8837393 | Standard disease code |
| Coronary artery disease | 1200 | |

| Variable Used in Study | ICD-10<br>Code <sup>*</sup> | Additional rules on Data Extraction |
|---|---|---|
| | 1201 | |
| | 1208 | |
| | 1209 | |
| | I210 | |
| | I211 | |
| | 1212 | |
| | I213 | |
| | I214 | |
| | 1240 | |
| | 1241 | |
| | 1248 | |
| | I251 | |
| | 1252 | Exclude calcification of coronary artery |
| | 1255 | |
| | 1258 | Exclude coronary arteritis |
| | 1259 | |
| Myocardial infarction | 1200 | Exclude intermediate angina syndrome, preinfarction syndrome, initial arbeits angina, intermediate coronary syndrome |
| | I210 | - Cyriai onio |
| | I211 | |
| | 1212 | |
| | 1214 | |
| | 1240 | |
| | 1241 | Exclude Dressler syndrome |
| Renal impairment | l120 | |
| | I129 | |
| | I139 | |
| | N003 | |
| | N009 | |
| | N032 | |
| | N033 | |
| | N039 | |
| | N040 | |
| | N044 | |
| | N049 | |
| | N052 | |

ICD-10 Variable Used Additional rules Code\* in Study on Data Extraction N055 N058 N059 N170 N171 N172 N178 N179 N189 N19 Exclude renal anemia, afunctional kidney, and alimentary proteinuria Liver dysfunction B150 B159 B162 B169 B171 B172 B178 B179 B181 B182 B189 B190 B199 C220 K700 K701 K703 K709 K716 K720 K721 K729 K730 K732 K738 K739 K740

| Variable Used in Study | ICD-10<br>Code* | Additional rules on Data Extraction |
|---|---|---|
| iii Study | K741 | On Data Extraction |
| | K743 | |
| | K744 | |
| | K745 | |
| | K746 | |
| | K750 | |
| | K751 | |
| | K754 | |
| | K759 | |
| | K760 | |
| | K761 | |
| | K762 | |
| | K763 | |
| | K766 | |
| | K767 | |
| | K768 | |
| | K769 | |
| Cancer | C00 | |
| | C01 | |
| | C02 | |
| | C03 | |
| | C04 | |
| | C05 | |
| | C06 | |
| | C07 | |
| | C08 | |
| | C09 | |
| | C10 | |
| | C11 | |
| | C12 | |
| | C13 | |
| | C14 | |
| | C15 | |
| | C16 | |
| | C17 | |
| | C18 | |
| | C19 | |

| Variable Used in Study | ICD-10<br>Code* | Additional rules on Data Extraction |
|---|---|---|
| | C20 | |
| | C21 | |
| | C22 | |
| | C23 | |
| | C24 | |
| | C25 | |
| | C26 | |
| | C30 | |
| | C31 | |
| | C32 | |
| | C33 | |
| | C34 | |
| | C37 | |
| | C38 | |
| | C40 | |
| | C41 | |
| | C43 | |
| | C44 | |
| | C45 | |
| | C46 | |
| | C47 | |
| | C48 | |
| | C49 | |
| | C50 | |
| | C51 | |
| | C52 | |
| | C53 | |
| | C54 | |
| | C55 | |
| | C56 | |
| | C57 | |
| | C58 | |
| | C60 | |
| | C61 | |
| | C62 | |
| | C63 | |

ICD-10 Variable Used Additional rules Code\* in Study on Data Extraction C64 C65 C66 C67 C68 C69 C70 C71 C72 C73 C74 C75 C76 C78 C79 C80 C81 C82 C83 C84 C85 C88 C90 C91 C92 C93 C94 C95 C96 C97 D00 D01 D02 D03 D04 D05

ICD-10 Variable Used Additional rules in Study Code\* on Data Extraction D06 D07 D09 D10 D11 D12 D13 D14 D15 D16 D17 D18 D19 D20 D21 D22 D23 D24 D25 D27 D28 D29

# PFIZER CONFIDENTIAL

D30
D31
D32
D33
D34
D35
D36
D37
D38
D39
D40
D41
D42
D43

 Variable Used in Study
 ICD-10 Code\*
 Additional rules on Data Extraction

 D44
 D45

 D46
 D48

# 10.3.2. List of procedure code

| Procedure | Procedure Code |
|-----------------|----------------|
| Cardiac surgery | 150138210 |
| | 150138310 |
| | 150138410 |
| | 150138510 |
| | 150359210 |
| | 150138710 |
| | 150140510 |
| | 150140610 |
| | 150140710 |
| | 150139010 |
| | 150140810 |
| | 150318010 |
| | 150317810 |
| | 150318110 |
| | 150331450 |
| | 150331550 |
| | 150331950 |
| | 150332050 |
| | 150317910 |
| | 150318210 |
| | 150140010 |
| | 150139210 |
| | 150153910 |
| | 150374910 |
| | 150375010 |
| | 150375110 |
| | 150260350 |
| | 150284310 |
| | 150359310 |
| | 150263310 |

| Procedure | Procedure Code |
|-----------|----------------|
| | 150375210 |
| | 150375310 |
| | 150375410 |
| | 160107550 |
| | 150139810 |
| | 150139910 |
| | 150318310 |
| | 150145710 |
| | 150145810 |
| | 150145910 |
| | 150146010 |
| | 150318410 |
| | 150318510 |
| | 150302770 |
| | 150143010 |
| | 150143110 |
| | 150331650 |
| | 150332150 |
| | 150318710 |
| | 150319010 |
| | 150319310 |
| | 150318810 |
| | 150319110 |
| | 150319410 |
| | 150328750 |
| | 150328850 |
| | 150331750 |
| | 150331850 |
| | 150332250 |
| | 150332350 |
| | 150318910 |
| | 150319210 |
| | 150319510 |
| | 150318610 |
| | 150141010 |
| | 150279510 |
| | 150279610 |
| | 150141410 |

| Procedure | Procedure Code |
|-----------|----------------|
| | 150141610 |
| | 150369950 |
| | 150141710 |
| | 150359470 |
| | 150143610 |
| | 150260050 |
| | 150143710 |
| | 150143810 |
| | 150141510 |
| | 150375570 |
| | 150375670 |
| | 150375770 |
| | 150319610 |
| | 150292910 |
| | 150139310 |
| | 150140910 |
| | 150242550 |
| | 150244910 |
| | 150245010 |
| | 150359510 |
| | 150359610 |
| | 150381150 |
| | 150381250 |
| | 150381350 |
| | 150381450 |
| | 150150010 |
| | 150381550 |
| | 150275910 |
| | 150359710 |
| | 150359810 |
| | 150359910 |
| | 150381650 |
| | 150381750 |
| | 150381850 |
| | 150381950 |
| | 150150110 |
| | 150382050 |
| | 150245110 |

| Procedure | Procedure Code |
|-----------|----------------|
| | 150245210 |
| | 150375870 |
| | 150375970 |
| | 150376070 |
| | 150141210 |
| | 150301310 |
| | 150267850 |
| | 150319710 |
| | 150151810 |
| | 150376110 |
| | 150139110 |
| | 150319810 |
| | 150138810 |
| | 150151910 |
| | 150320010 |
| | 150346410 |
| | 150320110 |
| | 150147150 |
| | 150144110 |
| | 150320210 |
| | 150320310 |
| | 150142710 |
| | 150139410 |
| | 150320410 |
| | 150142910 |
| | 150320510 |
| | 150260150 |
| | 150346510 |
| | 150145110 |
| | 150145010 |
| | 150376210 |
| | 150376310 |
| | 150143250 |
| | 150143350 |
| | 150143450 |
| | 150143550 |
| | 150283250 |
| | 150283350 |

| Procedure | Procedure Code |
|-----------|----------------|
| | 150283450 |
| | 150283550 |
| | 150144910 |
| | 150139610 |
| | 150142410 |
| | 150141810 |
| | 150141910 |
| | 150320610 |
| | 150142050 |
| | 150142110 |
| | 150142210 |
| | 150142310 |
| | 150142810 |
| | 150144010 |
| | 150320710 |
| | 150144210 |
| | 150144550 |
| | 150147410 |
| | 150147510 |
| | 150320810 |
| | 150320910 |
| | 150144410 |
| | 150144650 |
| | 150144750 |
| | 150146510 |
| | 150146610 |
| | 150321010 |
| | 150321110 |
| | 150321210 |
| | 150376470 |
| | 150146910 |
| | 150146810 |
| | 150321310 |
| | 150142510 |
| | 150329810 |
| | 150145310 |
| | 150329910 |
| | 150139510 |
NIS Protocol <B0661181>

| Procedure | Procedure Code |
|-----------|----------------|
| | 150330010 |
| | 150147010 |
| | 150330110 |
| | 150376570 |
| | 150321410 |
| | 150321510 |
| | 150376670 |
| | 150147310 |
| | 150145650 |
| | 150141310 |
| | 150321810 |
| | 150321610 |
| | 150321910 |
| | 150146710 |
| | 150321710 |
| | 150330210 |
| | 150330310 |
| | 150376770 |
| | 150293010 |
| | 150330410 |
| | 150145510 |
| | 150302870 |
| | 150145410 |
| | 150322010 |
| | 150322110 |
| | 150144310 |
| | 150147250 |
| | 150346610 |
| | 150144810 |
| | 150253810 |
| | 150253910 |
| | 150275610 |
| | 150346710 |
| | 150262810 |
| | 150303310 |
| | 150267310 |
| | 150140110 |
| | 150140210 |


| Procedure | Procedure Code |
|-----------|----------------|
| | 150140410 |
| | 150346910 |
| | 150347010 |
| | 150303210 |
| | 150322210 |
| | 150275210 |
| | 150275310 |
| | 150336910 |
| | 150337010 |
| | 150360010 |
| | 150148010 |
| | 150148110 |
| | 150147610 |
| | 150147910 |
| | 150147770 |
| | 150147870 |
| | 150347170 |
| | 150275870 |
| | 150262910 |
| | 150275710 |
| | 150266110 |
| | 150382650 |
| | 150266210 |
| | 150382750 |
| | 150301810 |
| | 150382850 |
| | 150303410 |
| | 150303510 |
| | 150360110 |
| | 150360210 |
| | 150360310 |
| | 150360410 |
| | 150303610 |
| | 150303710 |
| | 150322410 |
| | 150322610 |
| Ablation | 150346710 |
| | 150262810 |

## PFIZER CONFIDENTIAL

| Procedure | Procedure Code |
|---------------------------------------------|----------------|
| | 150303310 |
| | 150346870 |
| | 150370050 |
| Electrical defibrillation | 140051410 |
| | 140010310 |
| | 140055010 |
| | 150275210 |
| | 150275310 |
| | 150336910 |
| | 150337010 |
| | 150370550 |
| Heart valve prosthesis implantation surgery | 150141410 |
| | 150141610 |
| | 150141710 |
| | 150359470 |
| | 150369950 |
| | 150331950 |
| | 150332050 |
| | 150332150 |
| | 150328850 |
| | 150332250 |
| | 150332350 |
| | 150141510 |
| | 150375570 |
| | 150375670 |
| | 150375770 |
| | 150244910 |
| | 150359510 |
| | 150381150 |
| | 150381250 |
| | 150359710 |
| | 150359810 |
| | 150381650 |
| | 150381750 |
| | 150283450 |

## 10.3.3. Stroke related medical history

| Disease | ICD10<br>code | Standard<br>disease<br>code | Note |
|---|---|---|---|
| Homorrhogo | 160 | | |
| Hemorrhage<br>stroke | l61 | | |
| Sti Oke | 162 | | Exclude non-traumatic extradural haemorrhage |
| | 163 | | |
| | - | 3489032 | |
| | - | 4371003 | |
| | | 4379014 | |
| Ischemic stroke | | 3448002 | |
| | | 3448028 | |
| | | 3489029 | |
| | | 3489035 | |
| | | 4379006 | |
| | H340 | | |
| | G450 | | |
| TIA | G451 | | |
| | G458 | | |
| | G459 | | |
| | 1740 | | Include only abdominal aortic embolism |
| | 1741 | | Include only aortic embolism |
| | 1742 | | Include only acute arterial occlusive disease of arteries of upper extremities |
| Systemic | 1743 | | Include only femoral arterial occlusion and acute arterial occlusive disease of arteries of lower extremities |
| embolism | 1744 | | |
| | 1745 | | Include only iliac artery embolism |
| | 1748 | | Include only hepatic artery embolism |
| | 1749 | | Include only thromboembolism, embolic infarction, aortic embolism |
| | 1748 | | Include only subclavian artery stenosis |

## 10.3.4. bleeding

Procedure for definition of "bleeding"

Step 1. To extract the following group A or group B from MDV data base.

Group A: ICD-10 name includes "出血 (bleeding)" or "血腫 (ecchymoma)"

Group B: Disease name includes "出血 (bleeding)" or "血腫 (ecchymoma)"

Step 2. To select disease names considered to be relevant to side effect of OAC individually from disease names excluded in Step 1.

Step 3. To exclude disease names which are not considered to be relevant to side effect of OAC from the disease names included in Step 1.

| ICD-10 | ICD10Name |
|---|---|
| A162 | Tuberculosis of lung, without mention of bacteriological or histological confirmation |
| A165 | Tuberculous pleurisy, without mention of bacteriological or histological confirmation |


| ICD-10 | ICD10Name |
|---|---|
| B303 | Acute epidemic haemorrhagic conjunctivitis (enteroviral) |
| D500 | Iron deficiency anaemia secondary to blood loss (chronic) |
| D62 | Acute posthaemorrhagic anaemia |
| D66 | Hereditary factor VIII deficiency |
| D683 | Haemorrhagic disorder due to circulating anticoagulants |
| D698 | Other specified haemorrhagic conditions |
| D699 | Haemorrhagic condition, unspecified |
| E078 | Other specified disorders of thyroid |
| E274 | Other and unspecified adrenocortical insufficiency |
| G361 | Acute and subacute haemorrhagic leukoencephalitis [Hurst] |
| G951 | Vascular myelopathies |
| G968 | Other specified disorders of central nervous system |
| H052 | Exophthalmic conditions |
| H113 | Conjunctival haemorrhage |
| H168 | Other keratitis |
| H208 | Other iridocyclitis |
| H210 | Hyphaema |
| H313 | Choroidal haemorrhage and rupture |
| H350 | Background retinopathy and retinal vascular changes |
| H356 | Retinal haemorrhage |
| H357 | Separation of retinal layers |
| H405 | Glaucoma secondary to other eye disorders |
| H431 | Vitreous haemorrhage |
| H448 | Other disorders of globe |
| H470 | Disorders of optic nerve, not elsewhere classified |
| H603 | Other infective otitis externa |
| H669 | Otitis media, unspecified |
| H738 | Other specified disorders of tympanic membrane |
| H922 | Otorrhagia |
| I213 | Acute transmural myocardial infarction of unspecified site |
| 1230 | Haemopericardium as current complication following acute myocardial infarction |
| I312 | Haemopericardium, not elsewhere classified |
| 1600 | Subarachnoid haemorrhage from carotid siphon and bifurcation |
| I601 | Subarachnoid haemorrhage from middle cerebral artery |
| 1602 | Subarachnoid haemorrhage from anterior communicating artery |
| 1603 | Subarachnoid haemorrhage from posterior communicating artery |
| 1604 | Subarachnoid haemorrhage from basilar artery |
| 1605 | Subarachnoid haemorrhage from vertebral artery |
| 1606 | Subarachnoid haemorrhage from other intracranial arteries |
| 1607 | Subarachnoid haemorrhage from intracranial artery, unspecified |
| 1608 | Other subarachnoid haemorrhage |
| 1609 | Subarachnoid haemorrhage, unspecified |

ICD-10 ICD10Name 1610 Intracerebral haemorrhage in hemisphere, subcortical 1611 Intracerebral haemorrhage in hemisphere, cortical 1613 Intracerebral haemorrhage in brain stem 1614 Intracerebral haemorrhage in cerebellum 1615 Intracerebral haemorrhage, intraventricular 1616 Intracerebral haemorrhage, multiple localized 1618 Other intracerebral haemorrhage 1619 Intracerebral haemorrhage, unspecified 1620 Subdural haemorrhage (acute)(nontraumatic) 1621 Nontraumatic extradural haemorrhage 1629 Intracranial haemorrhage (nontraumatic), unspecified 1638 Other cerebral infarction 1690 Sequelae of subarachnoid haemorrhage 1691 Sequelae of intracerebral haemorrhage 1780 Hereditary haemorrhagic telangiectasia 1788 Other diseases of capillaries 1841 Internal hemorrhoid with other complications 1844 External hemorrhoid with other complications 1848 Unspecified hemorrhoid with other complications 1850 Oesophageal varices with bleeding 1864 Gastric varices J041 Acute tracheitis J339 Nasal polyp, unspecified J90 Pleural effusion, not elsewhere classified J942 Haemothorax J950 Tracheostomy malfunction K049 Other and unspecified diseases of pulp and periapical tissues K068 Other specified disorders of gingiva and edentulous alveolar ridge K121 Other forms of stomatitis K137 Other and unspecified lesions of oral mucosa K148 Other diseases of tongue K226 Gastro-oesophageal laceration-haemorrhage syndrome K228 Other specified diseases of oesophagus K250 Acute with haemorrhage K252 Gastric ulcer, Acute with both haemorrhage and perforation K254 Gastric ulcer, Chronic or unspecified with haemorrhage K256 Gastric ulcer, Chronic or unspecified with both haemorrhage and perforation K260 Duodenal ulcer, Acute with haemorrhage Duodenal ulcer, Acute with both haemorrhage and perforation K262 K264 Duodenal ulcer, Chronic or unspecified with haemorrhage K266 Duodenal ulcer, Chronic or unspecified with both haemorrhage and perforation K270 Acute duodenal tumor with haemorrhage

ICD-10 ICD10Name Gastrojejunal ulcer, Chronic or unspecified with haemorrhage K284 K290 Acute haemorrhagic gastritis K571 Diverticular disease of small intestine without perforation or abscess K573 Diverticular disease of large intestine without perforation or abscess K625 Haemorrhage of anus and rectum K661 Haemoperitoneum K762 Central haemorrhagic necrosis of liver K768 Other specified diseases of liver K85 Acute pancreatitis K920 Haematemesis K921 Melaena K922 Gastrointestinal haemorrhage, unspecified L508 Other urticaria M250 Haemarthrosis N029 Recurrent and persistent haematuria, Unspecified N288 Other specified disorders of kidney and ureter N300 Acute cystitis N304 Irradiation cystitis N309 Cystitis, unspecified N328 Other specified disorders of bladder N368 Other specified disorders of urethra N421 Congestion and haemorrhage of prostate N488 Other specified disorders of penis N501 Vascular disorders of male genital organs N645 Other signs and symptoms in breast N830 Follicular cyst of ovary N831 Corpus luteum cyst N836 Haematosalpinx N837 Haematoma of broad ligament N838 Other noninflammatory disorders of ovary, fallopian tube and broad ligament N898 Other specified noninflammatory disorders of vagina N908 Other specified noninflammatory disorders of vulva and perineum N921 Excessive and frequent menstruation with irregular cycle N922 Excessive menstruation at puberty N923 Ovulation bleeding N924 Excessive bleeding in the premenopausal period N930 Postcoital and contact bleeding N938 Other specified abnormal uterine and vaginal bleeding N939 Abnormal uterine and vaginal bleeding, unspecified N950 Postmenopausal bleeding O208 Other haemorrhage in early pregnancy O209 Haemorrhage in early pregnancy, unspecified

R195

R233

R31

ICD-10 ICD10Name O441 Placenta praevia with haemorrhage O469 Antepartum haemorrhage, unspecified O679 Intrapartum haemorrhage, unspecified O695 Labour and delivery complicated by vascular lesion of cord 0717 Obstetric haematoma of pelvis 0720 Third-stage haemorrhage 0721 Other immediate postpartum haemorrhage 0722 Delayed and secondary postpartum haemorrhage O901 Disruption of perineal obstetric wound O902 Haematoma of obstetric wound P021 Fetus and newborn affected by other forms of placental separation and haemorrhage P100 Subdural haemorrhage due to birth injury P101 Cerebral haemorrhage due to birth injury P102 Intraventricular haemorrhage due to birth injury Subarachnoid haemorrhage due to birth injury P103 P109 Unspecified intracranial laceration and haemorrhage due to birth injury P120 Cephalhaematoma due to birth injury P269 Unspecified pulmonary haemorrhage originating in the perinatal period P510 Massive umbilical haemorrhage of newborn P519 Umbilical haemorrhage of newborn, unspecified P523 Unspecified intraventricular (nontraumatic) haemorrhage of fetus and newborn P524 Intracerebral (nontraumatic) haemorrhage of fetus and newborn P528 Other intracranial (nontraumatic) haemorrhages of fetus and newborn P529 Intracranial (nontraumatic) haemorrhage of fetus and newborn, unspecified P540 Neonatal haematemesis P542 Neonatal rectal haemorrhage P543 Other neonatal gastrointestinal haemorrhage P544 Neonatal adrenal haemorrhage P545 Neonatal cutaneous haemorrhage P546 Neonatal vaginal haemorrhage P549 Neonatal haemorrhage, unspecified P580 Neonatal jaundice due to bruising P581 Neonatal jaundice due to bleeding R040 **Epistaxis** R041 Haemorrhage from throat R042 Haemoptysis R048 Haemorrhage from other sites in respiratory passages R049 Haemorrhage from respiratory passages, unspecified R18 Ascites

Other faecal abnormalities

Spontaneous ecchymoses

Unspecified haematuria

| ICD-10 | ICD10Name |
|---|---|
| R571 | Hypovolaemic shock |
| R58 | Haemorrhage, not elsewhere classified |
| S000 | Superficial injury of scalp |
| S001 | Contusion of eyelid and periocular area |
| S002 | Other superficial injuries of eyelid and periocular area |
| S003 | Superficial injury of nose |
| S004 | Superficial injury of ear |
| S005 | Superficial injury of lip and oral cavity |
| S007 | Multiple superficial injuries of head |
| S008 | Superficial injury of other parts of head |
| S013 | Open wound of ear |
| S019 | Open wound of head, part unspecified |
| S050 | Injury of conjunctiva and corneal abrasion without mention of foreign body |
| S051 | Contusion of eyeball and orbital tissues |
| S063 | Focal brain injury |
| S064 | Epidural haemorrhage |
| S065 | Traumatic subdural haemorrhage |
| S066 | Traumatic subarachnoid haemorrhage |
| S068 | Other intracranial injuries |
| S098 | Other specified injuries of head |
| S100 | Contusion of throat |
| S101 | Other and unspecified superficial injuries of throat |
| S141 | Other and unspecified injuries of cervical spinal cord |
| S241 | Other and unspecified injuries of thoracic spinal cord |
| S271 | Traumatic haemothorax |
| S272 | Traumatic haemopneumothorax |
| S278 | Injury of other specified intrathoracic organs |
| S279 | Injury of unspecified intrathoracic organ |
| S301 | Contusion of abdominal wall |
| S302 | Contusion of external genital organs |
| S341 | Other injury of lumbar spinal cord |
| S361 | Injury of liver or gallbladder |
| S368 | Injury of other intra-abdominal organs |
| S369 | Injury of unspecified intra-abdominal organ |
| S370 | Injury of kidney |
| S378 | Injury of other pelvic organs |
| S390 | Injury of muscle and tendon of abdomen, lower back and pelvis |
| S400 | Contusion of shoulder and upper arm |
| S408 | Other superficial injuries of shoulder and upper arm |
| S500 | Contusion of elbow |
| S501 | Contusion of other and unspecified parts of forearm |
| S600 | Contusion of finger(s) without damage to nail |

ICD10Name ICD-10 S601 Contusion of finger(s) with damage to nail S701 Contusion of thigh S800 Contusion of knee S801 Contusion of other and unspecified parts of lower leg S901 Contusion of toe(s) without damage to nail S902 Contusion of toe(s) with damage to nail T009 Multiple superficial injuries, unspecified T060 Injuries of brain and cranial nerves with injuries of nerves and spinal cord at neck level T090 Superficial injury of trunk, level unspecified T093 Injury of spinal cord, level unspecified Superficial injury of unspecified body region T140 T144 Injury of nerve(s) of unspecified body region T145 Injury of blood vessel(s) of unspecified body region T146 Injury of muscles and tendons of unspecified body region T794 Traumatic shock T810 Haemorrhage and haematoma complicating a procedure, not elsewhere classified T811 Shock during or resulting from a procedure, not elsewhere classified T876 Other and unspecified complications of amputation stump T905 Sequelae of intracranial injury Subgaleal hemorrhage Intracranial hemorrhage

## 10.3.5. other codes

| Subgroups | ICD10<br>code | Standard<br>disease<br>code | Note |
|---|---|---|---|
| Hypertension | | | Refer to 10.3.1 |
| Liver dysfunction | | | Refer to 10.3.1 |
| Renal impairment | | | Refer to 10.3.1 |
| | A162 | | Include only tubercular hemoptysis |
| | A165 | | Include only tubercular hemothorax |
| | B303 | | |
| | D500 | | |
| | D62 | | |
| Bleeding | D66 | | Include only hemophiliac bleeding |
| history | D683 | | Include only hemorrhagic disorder due to circulating |
| | D003 | | anticoagulants |
| | D698 | | |
| | D699 | | |
| | E078 | | Include only thyroid bleeding |
| | E274 | | Include only adrenal bleeding |


| Subgroups | ICD10<br>code | Standard<br>disease<br>code | Note |
|---|---|---|---|
| | G361 | | |
| | | | Include only hematomyelia, spinal subdural |
| | G951 | | hemorrhage, hematorrhachis, spinal epidural |
| | 0001 | | hemorrhage and spontaneous Cervical Epidural |
| | | | Hematoma |
| | G968 | | Include only spinal subarachnoid hemorrhage |
| | H052 | | Include only orbital fat hemorrhage |
| | H113 | | Include only Homorrhogic Korotitie |
| | H168<br>H208 | | Include only Hemorrhagic keratitis |
| | H210 | | Include only hemorrhagic iritis |
| | H313 | | |
| | H350 | | Include only hemorrhagic retinitis and juvenile recurrent |
| | | | vitreoretinal hemorrhage |
| | H356 | | |
| | H357 | | Include only hemorrhagic retinal pigment epithelial detachment |
| | H405 | | Include only hemorrhagic glaucoma |
| | H431 | | |
| | H448 | | Include only intraocular hemorrhage |
| | H470 | | Include only optic disc hemorrhage and optic nerve sheath hemorrhage |
| | H603 | | Include only otitis externa hemorrhagica |
| | H669 | | Include only hemorrhagic otitis media |
| | H738 | | Include only eardrum bleeding |
| | H922 | | |
| | I213 | | Include only Atrial thrombus as current complication following acute myocardial infarction |
| | 1230 | | • |
| | I312 | | |
| | 1600 | | |
| | <u>1601</u> | | |
| | 1602 | | |
| | 1603 | | |
| | 1604 | | |
| | 1605 | | |
| | 1606 | | |
| | 1607 | | |
| | 1608 | | |
| | 1609 | | |
| | I610 | | |
| | 1611 | | |
| | I613 | | |
| | 1614<br>1615 | | |
| | 1616 | | |
| | 1618 | | |
| | 1010 | | |

| Subgroups | ICD10<br>code | Standard<br>disease<br>code | Note |
|---|---|---|---|
| | I619 | | |
| | 1620 | | |
| | l621 | | |
| | 1629 | | |
| | 1638 | | Include only hemorrhagic cerebral infarction |
| | 1690 | | |
| | 1691 | | |
| | 1780 | | |
| | 1788 | | |
| | 1850 | | |
| | 1864 | | Include only gastric variceal bleeding |
| | J041 | | Include only hemorrhagic tracheitis |
| | J339 | | Include only bleeding polyp |
| | J90 | | Include only hemorrhagic pleural effusion |
| | J942 | | |
| | J950 | | Include only bleeding from a tracheostomy site |
| | K049 | | Include only hemorrhage in the pulp |
| | K068 | | Include only gingival hemorrhage |
| | K121 | | Include only hemorrhagic stomatitis |
| | K137 | | Include only oral hemorrhage |
| | K148 | | Include only tongue root submucosal bleeding |
| | K226 | | |
| | K228 | | Include only esophageal hemorrhage |
| | K250 | | |
| | K252 | | |
| | K254 | | |
| | K256 | | |
| | K260 | | Exclude acute gastroduodenal mucosal lesion |
| | K262 | | |
| | K264 | | |
| | K266 | | |
| | K284 | | |
| | K290 | | |
| | K571 | | Include only Duodenal diverticulum bleeding |
| | K573 | | Include only bleeding from Sigmoid diverticulum, |
| | | | Transverse colon diverticulum, Descending colon |
| | | | diverticulum, Ascending colon diverticulum and Large intestine diverticulum |
| | K625 | | intestine diverticulum |
| | K649 | | Include only Hemorrhoidal external hemorrhoids, |
| | 11049 | | Hemorrhoids and Hemorrhoidal internal hemorrhoids |
| | K661 | | Homormolas and Homormoladi Internal Hemormolas |
| | K762 | | |
| | K768 | | Include only hepatorrhagia |
| | K859 | | Include only hepatormagia Include only acute hemorrhagic necrotizing pancreatitis |
| | K920 | | moduc only acute hemormagic necrotizing pancreatitis |
| | K920 | | |
| | 11921 | | |

| Subgroups | ICD10<br>code | Standard<br>disease<br>code | Note |
|---|---|---|---|
| | K922 | | |
| | L508 | | Include only hemorrhagic urticaria |
| | M2506 | | |
| | M2509 | | |
| | N029 | | |
| | N288 | | Include only perirenal bleeding, nephrorrhagia and idiopathic hematuria |
| | N300 | | Include only acute hemorrhagic cystitis |
| | N304 | | Include only radiation-induced hemorrhagic cystitis |
| | N309 | | Include only hemorrhagic cystitis |
| | N328 | | Include only bladder hemorrhage |
| | N368 | | Include only urethremorrhagia |
| | N421 | | |
| | N488 | | Include only penile hemorrhage |
| | N501 | | Include only Scrotal hemorrhage and Spermatic cord hematoma |
| | N645 | | Include only thelorrhagia |
| | N830 | | Include only follicular hemorrhage and hemorrhagic |
| | | | follicular cyst |
| | N831 | | Exclude luteal cyst |
| | N836 | | |
| | N837 | | |
| | N838 | | Include only ovarian hemorrhage |
| | N898 | | Include only vaginal hematoma |
| | N908 | | Include only vulval hemorrhage |
| | N921<br>N922 | | |
| | N922<br>N923 | | |
| | N923 | | |
| | N930 | | |
| | N938 | | |
| | N939 | | |
| | N950 | | |
| | 0717 | | |
| | O901 | | |
| | O902 | | |
| | R040 | | |
| | R041 | | |
| | R042 | | |
| | R048 | | |
| | R049 | | |
| | R18 | | Include only hemorrhagic ascites |
| | R195 | | Include only fecal occult blood |
| | R233 | | |
| | R31 | | |
| | R571 | | Include only hemorrhagic shock |
| _ | R58 | | |

| Subgroups | ICD10<br>code | Standard<br>disease<br>code | Note |
|---|---|---|---|
| | S000 | | Include only ecchymoma, hematoma and hemorrhage |
| | S001 | | Include only hematoma and hemorrhage |
| | S002 | | Include only hematoma |
| | S003 | | Include only hematoma and hemorrhage |
| | S004 | | Include only hematoma and hemorrhage |
| | S005 | | Include only hematoma and hemorrhage |
| | S007 | | Include only hematoma and hemorrhage |
| | S008 | | Include only hematoma |
| | S013 | | Include only hemorrhage |
| | S050 | | Include only Corneal hematoma |
| | S051 | | Include only traumatic vitreous hemorrhage and traumatic hyphema |
| | S063 | | Include only hematoma and hemorrhage |
| | S064 | | moduce only homatoma and homormage |
| | S065 | | |
| | S066 | | |
| | S068 | | Include only hematoma, hemorrhage |
| | S098 | | Include only hemorrhage |
| | S100 | | Include only hematoma |
| | S101 | | |
| | S141 | | Include only hematoma |
| | S241 | | Include only hematoma |
| | S271 | | |
| | S272 | | |
| | S278 | | Include only hematoma |
| | S279 | | Include only hematoma |
| | S301 | | Include only hematoma |
| | S302 | | Include only hematoma |
| | S341 | | Include only hematoma |
| | S361 | | Include only hematoma |
| | S368 | | Include only hemorrhage |
| | S369 | | Include only hematoma |
| | S370 | | Include only hematoma |
| | S378 | | Include only hemorrhage |
| | S390 | | Include only hematoma |
| | S400 | | Include only hematoma |
| | S408 | | Include only hematoma |
| | S500 | | Include only hematoma |
| | S501 | | Include only hematoma |
| | S600 | | Include only hematoma |
| | S601 | | Include only hematoma |
| | S701 | | Include only hematoma |
| | S800 | | Include only hematoma |
| | S801 | | Include only hematoma |
| | S902 | | Include only hematoma |
| | T009 | | Include only hematoma and hemorrage |
| | T060 | | Include only spinal subarachnoid hemorrhage |


| Subgroups | ICD10<br>code | Standard<br>disease<br>code | Note |
|---|---|---|---|
| | T090 | | Including only hematoma |
| | T093 | | Including only hematoma |
| | T140 | | Including only hematoma |
| | T144 | | Include only traumatic hematomyelia |
| | T145 | | Include only traumatic arterial hematoma |
| | T146 | | Include only Intramuscular hematoma |
| | T794 | | Include only traumatic hemorrhagic shock |
| | T810 | | Include only hematoma and hemorrage |
| | T811 | | Include only hemorragic shock |
| | T876 | | Include only hematoma |
| | T905 | | Include only sequelae after |
| Hemorrhage<br>stroke | | | Refer to 10.3.1 |
| Alcohol abuse | E244 | | |
| | E52 | | Include only Alcoholic pellagra |
| | F100 | | , , , , |
| | G312 | | |
| | G405 | | Include only alcoholic epilepsy |
| | G621 | | , |
| | G701 | | Include only alcoholic neuropathy |
| | G721 | | |
| | H470 | | Include only alcoholic optic neuropathy |
| | 1426 | | |
| | K292 | | |
| | K70 | | |
| | K852 | | |
| | K860 | | |
| | T519 | | |
| Antiplatelet drug | | | Refer to 5.4 |
| NSAIDs | | | Refer to 5.4 |
| Peptic ulcer | F54 | | Include only psychogenic gastric ulcer |
| | K221 | | |
| | K227 | | Include only Barrett's esophagus |
| | K25 | | |
| | K26 | | |
| | K27 | | |
| | K28 | | |
| | K51 | | |
| | K626 | | |
| | K633 | | |
| Active cancer | | | Refer to 10.3.1 |
| Diabetes mellitus | | | Refer to 10.3.1 |
| CCI | | | |
| | _ | | |